CLINICAL TRIAL: NCT01096056
Title: Safety and Immunogenicity of GSK2186877A Candidate Seasonal Influenza Vaccine in Healthy Children 6 to 35 Months of Age.
Brief Title: Trial to Evaluate the Safety and the Immunogenicity of GSK Biologicals' Influenza Vaccine GSK2186877A in Healthy Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 114182
Record Dates: First submitted 2010-03-29; First posted 2010-03-30 (Estimated); Results first posted 2012-05-10 (Estimated); Last update posted 2018-09-24 (Actual); Status verified 2016-09

CONDITIONS: Influenza
Keywords: Children; Influenza; Safety; Immunogenicity; Vaccine
MeSH Terms: conditions — Influenza, Human | interventions — fluarix

ARMS (2):
- Influenza vaccine GSK2186877A formulation 1 Group (Experimental): Subjects received 2 doses of influenza vaccine GSK2186877A formulation 1 at Day 0 and Day 21 and 1 dose of Fluarix vaccine at Month 6.
  Interventions: Biological: Influenza vaccine GSK2186877A formulation 1; Biological: Fluarix
- Influenza vaccine GSK2186877A formulation 2 Group (Experimental): Subjects received 1 dose of influenza vaccine GSK2186877A formulation 2 at Day 0 and 1 dose of Fluarix vaccine at Month 6.
  Interventions: Biological: Influenza vaccine GSK2186877A formulation 2; Biological: Fluarix

INTERVENTIONS:
Biological: Influenza vaccine GSK2186877A formulation 1 — Intramuscular administration, 2 doses
  Arms: Influenza vaccine GSK2186877A formulation 1 Group
Biological: Influenza vaccine GSK2186877A formulation 2 — Intramuscular administration, 1 dose
  Arms: Influenza vaccine GSK2186877A formulation 2 Group
Biological: Fluarix — Intramuscular administration, 1 dose

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of GlaxoSmithKline Biologicals' influenza vaccine GSK2186877A in healthy children 6 to 35 months of age.

This Protocol Posting has been updated following Amendment 1 of the Protocol, Jun 2010. The impacted sections are study design, outcome measures, intervention sections and number of subjects.

ELIGIBILITY:
Inclusion Criteria:

All subjects must satisfy ALL the following criteria at study entry:

* Subjects who the investigator believes that parent(s)/Legally Acceptable Representative(s) [LAR(s)] can and will comply with the requirements of the protocol.
* Children, male or female between, and including, 6 and 35 months of age at the time of the first vaccination.
* Written informed consent obtained from the parent(s)/LAR(s) of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Age appropriate scheduled childhood vaccinations completed to the best of parent(s)/LAR(s) knowledge.

Exclusion Criteria:

The following criteria should be checked at the time of study entry. If ANY exclusion criterion applies, the subject must not be included in the study:

* Child in care
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Prior receipt of any influenza vaccination (seasonal or pandemic) or planned administration during the study period.
* Planned administration of any vaccine 30 days prior and 30 days after any study vaccine administration.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose. For corticosteroids, this will mean prednisone >0.5 mg/kg of body weight, or equivalent. Inhaled and topical steroids are allowed.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* A family history of congenital or hereditary immunodeficiency.
* Any known or suspected allergy to any constituent of influenza or routine paediatric vaccines, a history of severe adverse reaction to any previous vaccination; or a history of anaphylactic-type reaction to consumption of egg proteins.
* History of any neurological disorders or seizures (including febrile convulsion).
* Acute or chronic, clinically-significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by medical history or physical examination.
* Acute disease and/or fever at the time of enrolment:

  * Fever is defined as temperature >= 37.5°C on oral, axillary or tympanic setting, or >=38.0°C on rectal setting.
  * Subjects with a minor illness (such as mild diarrhoea, mild upper respiratory infection) without fever might be enrolled at the discretion of the investigator.
* Administration of immunoglobulins and/or any blood products within the 3 month preceding the first dose of study vaccine or planned administration during the study period.
* Any condition which, in the opinion of the investigator, render the subject unfit for participation in the study.

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2010-04-05; Primary Completion 2010-12-13 (Actual); Study Completion 2010-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Seville, Spain

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 114182 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114182 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114182 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114182 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114182 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114182 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Influenza Vaccine GSK2186877A Formulation 1 Group: Subjects aged 6 to 35 months received 2 doses of new generation influenza vaccine GSK2186877A formulation 1 at Day 0 and Day 21 and 1 dose of Fluarix vaccine at Month 6.
- Influenza Vaccine GSK2186877A Formulation 2 Group: Subjects aged 6 to 35 months received 1 dose of new generation influenza vaccine GSK2186877A formulation 2 at Day 0 and 1 dose of Fluarix vaccine at Month 6.
Period: Overall Study
Arm/Group | Influenza Vaccine GSK2186877A Formulation 1 Group | Influenza Vaccine GSK2186877A Formulation 2 Group
Started | 20 | 20
Completed at Day 42 | 20 | 20
Completed | 20 | 19
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Influenza Vaccine GSK2186877A Formulation 1 Group | Influenza Vaccine GSK2186877A Formulation 2 Group | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: Months] | 23.2 (9.82) | 18.6 (7.46) | 20.90 (8.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 18
  Male | 9 | 13 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Fever Grade 2 or Higher
Description: Fever grade greater than or equal to 2 i.e. ≥ 2 was defined as axillary temperature >38 degree centigrade (°C).
Time Frame: Within 7 days following any vaccination with New generation influenza vaccine GSK2186877A
Population: The analysis was performed on Total Vaccinated cohort which included all subjects with the vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza Vaccine GSK2186877A Formulation 1 Group | Influenza Vaccine GSK2186877A Formulation 2 Group
Number analyzed (Participants) | 20 | 20
Participants | 11 | 7

2. Secondary Outcome: Haemagglutination Inhibition (HI) Antibody Titers
Description: Antibody titers were expressed as Geometric mean titers (GMTs). The vaccine strains included Flu A/CAL/7/09 H1N1, Flu A/Uru/716/07 H3N2 and FluB/Bri/60/08 Victoria antigens.
Time Frame: At Day 0 and Day 42
Population: The immunogenicity analysis was based on the Total Vaccinated cohort which included all vaccinated subjects for whom immunogenicity data were available.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Influenza Vaccine GSK2186877A Formulation 1 Group | Influenza Vaccine GSK2186877A Formulation 2 Group
Number analyzed (Participants) | 20 | 20
Titers
  Flu A/CAL/7/09 H1N1 strain at Day 0 | 13.7 [6.5 to 28.9] | 35.4 [13.6 to 92.6]
  Flu A/CAL/7/09 H1N1 strain at Day 42: number analyzed (Participants) | 20 | 19
  Flu A/CAL/7/09 H1N1 strain at Day 42 | 905.2 [649.0 to 1262.6] | 617.1 [251.0 to 1516.8]
  Flu A/Uru/716/07 H3N2 strain at Day 0 | 14.9 [6.6 to 33.5] | 7.6 [4.1 to 13.9]
  Flu A/Uru/716/07 H3N2 strain at Day 42: number analyzed (Participants) | 20 | 19
  Flu A/Uru/716/07 H3N2 strain at Day 42 | 722.5 [473.8 to 1101.7] | 160.0 [86.3 to 296.7]
  FluB/Bri/60/08 Victoria strain at Day 0 | 5.9 [4.1 to 8.5] | 5.9 [4.1 to 8.5]
  FluB/Bri/60/08 Victoria strain at Day 42: number analyzed (Participants) | 20 | 19
  FluB/Bri/60/08 Victoria strain at Day 42 | 460.5 [320.4 to 661.8] | 63.1 [30.9 to 128.8]

3. Secondary Outcome: The Number of Subjects Seropositive to HI Antibodies
Description: A seropositive subject was defined as a subject with antibody titer greater than or equal to 1:10. The vaccine strains included Flu A/CAL/7/09 H1N1, Flu A/Uru/716/07 H3N2 and FluB/Bri/60/08 Victoria antigens.
Time Frame: At Day 0 and Day 42
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza Vaccine GSK2186877A Formulation 1 Group | Influenza Vaccine GSK2186877A Formulation 2 Group
Number analyzed (Participants) | 20 | 20
Participants
  Flu A/CAL/7/09 H1N1 strain at Day 0 | 6 | 10
  Flu A/CAL/7/09 H1N1 strain at Day 42: number analyzed (Participants) | 20 | 19
  Flu A/CAL/7/09 H1N1 strain at Day 42 | 20 | 19
  Flu A/Uru/716/07 H3N2 strain at Day 0 | 6 | 2
  Flu A/Uru/716/07 H3N2 strain at Day 42: number analyzed (Participants) | 20 | 19
  Flu A/Uru/716/07 H3N2 strain at Day 42 | 20 | 19
  FluB/Bri/60/08 Victoria strain at Day 0 | 1 | 1
  FluB/Bri/60/08 Victoria strain at Day 42: number analyzed (Participants) | 20 | 19
  FluB/Bri/60/08 Victoria strain at Day 42 | 20 | 19

4. Secondary Outcome: The Number of Subjects Seroprotected to HI Antibodies
Description: A seroprotected subject was defined as a subject with a serum HI titre greater than or equal to 1:40 that usually is accepted as indicating protection. The vaccine strains included Flu A/CAL/7/09 H1N1, Flu A/Uru/716/07 H3N2 and FluB/Bri/60/08 Victoria antigens.
Time Frame: At Day 0 and Day 42
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza Vaccine GSK2186877A Formulation 1 Group | Influenza Vaccine GSK2186877A Formulation 2 Group
Number analyzed (Participants) | 20 | 20
Participants
  Flu A/CAL/7/09 H1N1 strain at Day 0 | 6 | 10
  Flu A/CAL/7/09 H1N1 strain at Day 42: number analyzed (Participants) | 20 | 19
  Flu A/CAL/7/09 H1N1 strain at Day 42 | 20 | 19
  Flu A/Uru/716/07 H3N2 strain at Day 0 | 6 | 2
  Flu A/Uru/716/07 H3N2 strain at Day 42: number analyzed (Participants) | 20 | 19
  Flu A/Uru/716/07 H3N2 strain at Day 42 | 20 | 19
  FluB/Bri/60/08 Victoria strain at Day 0 | 1 | 1
  FluB/Bri/60/08 Victoria strain at Day 42: number analyzed (Participants) | 20 | 19
  FluB/Bri/60/08 Victoria strain at Day 42 | 20 | 14

5. Secondary Outcome: The Number of Subjects Seroconverted to HI Antibodies
Description: A seroconverted subject was defined as a subject who had either a pre-vaccination titer below 1:10 and a post-vaccination titer greater than or equal to 1:40 or a pre-vaccination titer greater than or equal to 1:10 and at least a 4-fold increase in post-vaccination titer. The vaccine strains included Flu A/CAL/7/09 H1N1, Flu A/Uru/716/07 H3N2 and FluB/Bri/60/08 Victoria antigens.
Time Frame: Day 42
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza Vaccine GSK2186877A Formulation 1 Group | Influenza Vaccine GSK2186877A Formulation 2 Group
Number analyzed (Participants) | 20 | 19
Participants
  Flu A/CAL/7/09 H1N1 strain | 20 | 19
  Flu A/Uru/716/07 H3N2 strain | 20 | 19
  FluB/Bri/60/08 Victoria strain | 20 | 14

6. Secondary Outcome: HI Antibody Geometric Mean Fold Rise (GMFR)
Description: GMFR was defined as the fold increase in serum HI GMTs post-vaccination compared to pre-vaccination. The vaccine strains included Flu A/CAL/7/09 H1N1, Flu A/Uru/716/07 H3N2 and FluB/Bri/60/08 Victoria antigens.
Time Frame: Day 42
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Influenza Vaccine GSK2186877A Formulation 1 Group | Influenza Vaccine GSK2186877A Formulation 2 Group
Number analyzed (Participants) | 20 | 19
fold change
  Flu A/CAL/7/09 H1N1 strain | 66.3 [38.8 to 113.3] | 19.6 [13.4 to 28.5]
  Flu A/Uru/716/07 H3N2 strain | 48.5 [28.0 to 84.1] | 20.7 [14.8 to 28.8]
  FluB/Bri/60/08 Victoria strain | 77.4 [59.4 to 101.0] | 10.5 [6.3 to 17.6]

7. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Adverse Events (AEs)
Description: Grade 3 redness and swelling was > 50 millimeter (mm) and grade 3 pain was subjects crying when limb was moved/spontaneously painful. Any was occurrence of any local symptom regardless of their intensity grade.
Time Frame: Within 7 days following any vaccination with New generation influenza vaccine GSK2186877A
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza Vaccine GSK2186877A Formulation 1 Group | Influenza Vaccine GSK2186877A Formulation 2 Group
Number analyzed (Participants) | 20 | 20
Participants
  Any pain | 10 | 6
  Grade 3 pain | 0 | 0
  Any redness | 7 | 2
  Grade 3 redness | 0 | 0
  Any swelling | 6 | 1
  Grade 3 swelling | 0 | 0

8. Secondary Outcome: Duration of Solicited Local AEs
Description: Duration was defined as number of days with any grade of local symptoms following each dose of New generation influenza vaccine GSK2186877A. Dose 1 application of vaccine involved Influenza vaccine GSK2186877A formulation 1 Group and Influenza vaccine GSK2186877A formulation 2 Group while Dose 2 involved only Influenza vaccine GSK2186877A formulation 1 Group.
Time Frame: Within 7 days following any vaccination with New generation influenza vaccine GSK2186877A
Population: The analysis was performed on Total Vaccinated cohort which included all subjects with the vaccine administration documented and symptom sheet completed only on subjects that reported the specific symptom.
Measure: Median (Full Range); unit: Days
Arm/Group | Influenza Vaccine GSK2186877A Formulation 1 Group | Influenza Vaccine GSK2186877A Formulation 2 Group
Number analyzed (Participants) | 7 | 6
Days
  Pain [Dose 1]: number analyzed (Participants) | 6 | 6
  Pain [Dose 1] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Pain [Dose 2] | 2.0 [1.0 to 2.0] | NA [NA to NA] — Subjects did not receive any second vaccine dose, as per protocol.
  Redness [Dose 1]: number analyzed (Participants) | 2 | 2
  Redness [Dose 1] | 3.5 [2.0 to 5.0] | 1.0 [1.0 to 1.0]
  Redness [Dose 2]: number analyzed (Participants) | 6 | 6
  Redness [Dose 2] | 2.5 [2.0 to 3.0] | NA [NA to NA] — Subjects did not receive any second vaccine dose, as per protocol.
  Swelling [Dose 1]: number analyzed (Participants) | 1 | 1
  Swelling [Dose 1] | 3.0 [3.0 to 3.0] | 1.0 [1.0 to 1.0]
  Swelling [Dose 2]: number analyzed (Participants) | 5 | 6
  Swelling [Dose 2] | 3.0 [2.0 to 4.0] | NA [NA to NA] — Subjects did not receive any second vaccine dose, as per protocol.

9. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General AEs
Description: Any temperature was defined as axillary temperature ≥37.5°C, grade 3 temperature was axillary temperature >39.0°C. For other symptoms, any was defined as occurrence of any symptom regardless of intensity grade or relation to vaccination. Grade 3 drowsiness was defined as general symptom that prevented normal activity, grade 3 irritability was crying that cannot be comforted/prevented normal activity, grade 3 loss of appetite was not eating at all and grade 3 vomiting was defined as ≥3 episode of vomiting/day. Related was symptom assessed by the investigator as causally related to vaccination.
Time Frame: Within 7 days following any vaccination with New generation influenza vaccine GSK2186877A
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza Vaccine GSK2186877A Formulation 1 Group | Influenza Vaccine GSK2186877A Formulation 2 Group
Number analyzed (Participants) | 20 | 20
Participants
  Any drowsiness | 6 | 7
  Grade 3 drowsiness | 0 | 1
  Related drowsiness | 3 | 3
  Any irritability | 7 | 9
  Grade 3 irritability | 1 | 1
  Related irritability | 4 | 4
  Any loss of appetite | 12 | 5
  Grade 3 loss of appetite | 0 | 1
  Related loss of appetite | 5 | 3
  Any temperature | 14 | 12
  Grade 3 temperature | 2 | 1
  Related temperature | 9 | 9
  Any vomiting | 7 | 4
  Grade 3 vomiting | 2 | 1
  Related vomiting | 2 | 0

10. Secondary Outcome: Duration of Solicited General AEs
Description: Duration was defined as number of days with any grade of local symptoms following each dose of New generation influenza vaccine GSK2186877A. Dose 1 application of vaccine involved subjects in Influenza vaccine GSK2186877A formulation 1 Group and Influenza vaccine GSK2186877A formulation 2 Group while Dose 2 application of vaccine involved only subjects in the Influenza vaccine GSK2186877A formulation 1 Group.
Time Frame: Within 7 days following any vaccination with New generation influenza vaccine GSK2186877A
Population: as for outcome 8
Measure: Median (Full Range); unit: Days
Arm/Group | Influenza Vaccine GSK2186877A Formulation 1 Group | Influenza Vaccine GSK2186877A Formulation 2 Group
Number analyzed (Participants) | 9 | 12
Days
  Drowsiness [Dose 1]: number analyzed (Participants) | 4 | 7
  Drowsiness [Dose 1] | 1.5 [1.0 to 3.0] | 2.0 [1.0 to 6.0]
  Drowsiness [Dose 2]: number analyzed (Participants) | 4 | 12
  Drowsiness [Dose 2] | 2.0 [1.0 to 4.0] | NA [NA to NA] — Subjects did not receive any second vaccine dose, as per protocol.
  Irritability [Dose 1]: number analyzed (Participants) | 4 | 9
  Irritability [Dose 1] | 2.5 [1.0 to 4.0] | 2.0 [1.0 to 6.0]
  Irritability [Dose 2]: number analyzed (Participants) | 4 | 12
  Irritability [Dose 2] | 1.0 [1.0 to 2.0] | NA [NA to NA] — Subjects did not receive any second vaccine dose, as per protocol.
  Loss of appetite [Dose 1]: number analyzed (Participants) | 9 | 5
  Loss of appetite [Dose 1] | 1.0 [1.0 to 3.0] | 2.0 [1.0 to 4.0]
  Loss of appetite [Dose 2]: number analyzed (Participants) | 5 | 12
  Loss of appetite [Dose 2] | 5.0 [1.0 to 6.0] | NA [NA to NA] — Subjects did not receive any second vaccine dose, as per protocol.
  Temperature [Dose 1]: number analyzed (Participants) | 7 | 12
  Temperature [Dose 1] | 1.0 [1.0 to 5.0] | 1.0 [1.0 to 6.0]
  Temperature [Dose 2] | 1.0 [1.0 to 4.0] | NA [NA to NA] — Subjects did not receive any second vaccine dose, as per protocol.
  Vomiting [Dose 1]: number analyzed (Participants) | 5 | 4
  Vomiting [Dose 1] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 2.0]
  Vomiting [Dose 2]: number analyzed (Participants) | 3 | 12
  Vomiting [Dose 2] | 1.0 [1.0 to 2.0] | NA [NA to NA] — Subjects did not receive any second vaccine dose, as per protocol.

11. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Unsolicited AEs
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as occurrence of any unsolicited symptom regardless of intensity grade or relation to vaccination. Grade 3 was event that prevented normal activities and Related was defined as unsolicited AE assessed by the investigator to be causally related to the study vaccination.
Time Frame: Within 21 days after any vaccination with New generation influenza vaccine GSK2186877A
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza Vaccine GSK2186877A Formulation 1 Group | Influenza Vaccine GSK2186877A Formulation 2 Group
Number analyzed (Participants) | 20 | 20
Participants
  Any AE(s) | 14 | 12
  Grade 3 AE(s) | 1 | 0
  Related AE(s) | 0 | 0

12. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related AEs With a Medically Attended Visit (MAEs)
Description: For each solicited and unsolicited AE the subject experienced, the subject was asked if they had received medical attention defined as hospitalization, an emergency room visit or a visit to or from medical personnel (medical doctor) for any reason. Any was defined as occurrence of any symptom regardless of intensity grade or relation to vaccination, grade 3 was defined as symptom that prevented normal activity and related was symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: Day 0 up to Month 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza Vaccine GSK2186877A Formulation 1 Group | Influenza Vaccine GSK2186877A Formulation 2 Group
Number analyzed (Participants) | 20 | 20
Participants
  Any MAE(s) | 18 | 20
  Grade 3 MAE(s) | 3 | 3
  Related MAE(s) | 0 | 0

13. Secondary Outcome: Number of Subjects Reporting Any Potential Immune-Mediated-Diseases (pIMDs)
Description: pIMDs are a subset of AEs that include both clearly autoimmune diseases and also other inflammatory and/or neurologic disorders which may or may not have an autoimmune etiology.
Time Frame: Day 0 up to Month 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza Vaccine GSK2186877A Formulation 1 Group | Influenza Vaccine GSK2186877A Formulation 2 Group
Number analyzed (Participants) | 20 | 20
Participants | 0 | 0

14. Secondary Outcome: Number of Subjects Reporting Any and Related Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject. Any was defined as occurrence of any symptom regardless of intensity grade or relation to vaccination and related was event assessed by the investigator as causally related to the study vaccination.
Time Frame: Day 0 up to Month 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza Vaccine GSK2186877A Formulation 1 Group | Influenza Vaccine GSK2186877A Formulation 2 Group
Number analyzed (Participants) | 20 | 20
Participants
  Any SAE (s) | 0 | 3
  Related SAE(s) | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events were assessed from day 0 up to month 7. Systematically assessed frequent adverse events (AEs) and Non-systematically assessed frequent AEs were assessed during 7 day and 21 day post vaccination period.
Arm/Group | Influenza Vaccine GSK2186877A Formulation 1 Group | Influenza Vaccine GSK2186877A Formulation 2 Group
Serious Adverse Events (participants affected / at risk) | 0/20 | 3/20
Other Adverse Events (participants affected / at risk) | 19/20 | 18/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Influenza Vaccine GSK2186877A Formulation 1 Group (N=20) | Influenza Vaccine GSK2186877A Formulation 2 Group (N=20)
Bronchopneumonia (Infections and infestations) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Influenza Vaccine GSK2186877A Formulation 1 Group (N=20) | Influenza Vaccine GSK2186877A Formulation 2 Group (N=20)
Pain (General disorders) | 10 | 6
Redness (General disorders) | 7 | 2
Swelling (General disorders) | 6 | 1
Drowsiness (General disorders) | 6 | 7
Irritability (General disorders) | 7 | 9
Loss of appetite (General disorders) | 12 | 5
Temperature (General disorders) | 14 | 12
Vomiting (General disorders) | 7 | 4
Upper respiratory tract infection (Infections and infestations) | 5 | 7
Pyrexia (General disorders) | 5 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Otitis media acute (Infections and infestations) | 3 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 | 2
Gastroenteritis (Infections and infestations) | 1 | 2
Nasopharyngitis (Infections and infestations) | 2 | 0
Teething (Gastrointestinal disorders) | 1 | 2
Conjunctivitis (Eye disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Haematoma (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.